CLINICAL TRIAL: NCT00972491
Title: The Optimal Time of Insertion of Laryngeal Mask Airway With Propofol Induction
Brief Title: The Optimal Time to Put Laryngeal Mask Airway in the Mouth Under General Anesthesia
Acronym: LMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-8910
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: General Anesthesia
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0 sec, 60 sec, 90 sec (Other): LMA will be inserted at 0, 60, and 90 seconds after eyelash reflex disappears
  Interventions: Procedure: Insertion of Laryngeal Mask Airway

INTERVENTIONS:
Procedure: Insertion of Laryngeal Mask Airway — The LMA will be inserted at 0 sec, 60 sec. and 90 sec. after induction of general anesthesia
  Other Names: Laryngeal Mask Airway

SUMMARY:
Laryngeal mask airway (LMA) is routinely used for some patients who have surgery under general anesthesia. LMA is placed in the mouth and allow the anesthesia to be given without having to put a breathing tube in the throat. Previous studies have focused on the effect of different anesthesia medicines on optimal condition for LMA use. The objective of the present study is to find the optimal time for LMA insertion.

DETAILED DESCRIPTION:
This is a randomized, controlled, blinded trial. Midazolam, 2 mg and fentanyl 1.0 µg/kg, would be given prior to induction with propofol, 2.5 mg/kg.

The investigator who does the induction of general anesthesia will also be responsible for the timekeeping. For this reason, it is not possible for this investigator to be blinded to randomization. The induction would conclude after loss of eyelash reflex (LER). At that point insertion of the LMA (#4 for females, #5 for males) will occur 0, 60 and 90 seconds after LER. The LMA will be lubricated with a water soluble gel and will be inserted with a deflated cuff according to the technique described by Brain.

The investigator who inserts the LMA (Inv1) will be in the operating room and blinded to randomization groups by not seeing the induction of general anesthesia. This investigator will insert the LMA only when called by the investigator who induces general anesthesia (Inv2). Inv1 will also grade ease of LMA insertion.

The primary outcome is Jaw opening at the time of LMA insertion, defined as full 1, partial 2, and nil 3.

Secondary outcomes include:

1. Insertion of LMA (easy, difficult, impossible)
2. Coughing or gagging (none, some, significant)
3. Head or body movement (none, some, significant)
4. Laryngospasm or airway obstruction (none, partial, total)

ELIGIBILITY:
Inclusion Criteria:

* subjects 18 years or older
* ASA status 1-3

Exclusion Criteria:

* high risk of aspiration
* anticipated difficult airway
* use of sedative drugs
* patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Ease of Mouth opening | From Induction of general anesthesia to satisfactory LMA insertion

CONTACTS AND LOCATIONS:
Overall Officials: Pei-shan Zhao, MD,PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States